CLINICAL TRIAL: NCT01230112
Title: TAP0307.6: Sub-study of TAP 0307- Enrollment of Normal Controls to Study the Role of ITGAM in Systemic Lupus Erythematosus
Brief Title: The Role of ITGAM in Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-289
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and DNA will be collected and retained
Oversight: Data Monitoring Committee: No

SUMMARY:
Study to examine the role of ITGAM molecule in normal control subjects with known genetic variation in the ITGAM gene.

ELIGIBILITY:
Inclusion Criteria:

* males and females, age 18 or older, enrolled in Genotype and Phenotype Registry, in general good health
* Participants who carry the genotype of interest, based on a buccal or blood derived DNA sample

Exclusion Criteria:

* History of Systemic Lupus Erythematosus, rheumatoid arthritis, or other autoimmune disease
* History of cancer or lymphoma
* Current use of aspirin, prednisone, or NSAID or any immunosuppressant
* Self reported HIV

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal Control Subjects with genotype of interest registered in the Genotype and Phenotype Registry
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States